CLINICAL TRIAL: NCT05224466
Title: Characteristics and Clinical Outcomes of Peritoneal Dialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Na Jiang, Associate Chief Physician of Nephrology, Shanghai Jiao Tong University School of Medicine
Other Study IDs: PD
Record Dates: First submitted 2021-12-14; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Peritoneal Dialysis Complication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- A: defined as patients survived on PD for more than 10 years
- B: defined as patients survived on PD for 5-10 years
- C: defined as patients survived on PD within 5 years

SUMMARY:
Peritoneal dialysis patients worldwide account for about 11% of the global dialysis population. The global annual growth rate of peritoneal dialysis is estimated to be 8%, which is listed as the preferred method of renal replacement therapy in most countries. Although peritoneal dialysis has been widely used, due to complications such as peritoneal dialysis related infection, peritoneal ultrafiltration failure and EPS, the failure rate of peritoneal dialysis technology is high, and the 3-year technical survival rate is only 64%. Therefore, this study intends to explore clinical strategies for maintaining the long-term peritoneal dialysis by analyzing the clinical characteristics of patients , as well as the differences of risk factors affecting the survival rate of peritoneal dialysis technology at different time stages of peritoneal dialysis treatment.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients
* The first time of peritoneal dialysis

Exclusion Criteria:

* Age <18 years at start of PD
* Transfer or follow-up loss
* Previous transplantation or HD history
* Incomplete clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ESRD patients who start the PD at the first time
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
baseline clinical characteristics before PD | within one month before the start of PD
  clinical characteristics about age,sex,comorbidities before PD,laboratory data would be aggregated from the existing record to find out the differences between the long-term PD patients and the others that may affect their clinical outcome.

SECONDARY OUTCOMES:
the factors that may lead to the termination of PD | up to 20 years
  Some patients may end the PD early ,some late due to many reasons.To find out the factors that may influence survival rate of peritoneal dialysis technology at different time stages of peritoneal dialysis treatment, the investigators collect and record the reasons for termination of PD to analyze.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Fang, MD, Study Director — RenJi Hospital
Locations (1):
- Shanghai Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No